CLINICAL TRIAL: NCT01748409
Title: Physiopathological Study of Autonomic Failure in Parkinson's Disease : a Monocentric Study
Brief Title: Physiopathological Study of Autonomic Failure in Parkinson's Disease
Acronym: SYNAPark
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RC12_0264
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Parkinson's Disease
Keywords: Autonomic failure, Parkinson's disease, electrophysiological assessment, neuropathological assessment
MeSH Terms: conditions — Parkinson Disease; Pure Autonomic Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Biopsies of peripheral autonomic nervous system
Other: Autonomic dysfunction questionnaires
  Other Names: a battery of questionaries to evaluate autonomic neurological patient complaints and dysfunctions.
Other: Electrophysiological tests
  Other Names: A battery of electrophysiological tests to assess neurological functions

SUMMARY:
The aim of the study is to evaluate the autonomic failure in Parkinson's disease by clinical, electrophysiological and neuropathological examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease
* ages 45 to 80 years, both genders
* patients who signed informed consent

Exclusion Criteria:

* autonomic function modifying treatment
* pre-existing neuropathy or risk factors for neuropathy
* dementia
* colonic disorders
* coagulation disorders (may be due to treatment)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Evaluate association between clinical autonomic failure and neuropathological autonomic failure on biopsies. | 3 months
  the main objective is to look after associations between :
  * anatomopathological signs of autonomic nervous system disorders seen on biopsies AND
  * clinical signs of signs of autonomic nervous system disorders seen through functional tests or through symptoms indicated by the patient on questionaries.

SECONDARY OUTCOMES:
Evaluate association between autonomic failure and severity factors in Parkinson's disease | 3 months
  Autonomic failure will be assessed through questionaries on symptoms and through functional tests.
  Severity factors in parkinson disease will refer to various parameters like patient age.
Evaluate consequences of autonomic failure on quality of life and sleep quality | 3 months
  quality of life and of sleep will be assessed through functional tests and through questionaries.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes Universitary Hospital, Nantes, Loire Atlantique, France

REFERENCES:
- [Derived] Sadoc M, Clairembault T, Coron E, Berthomier C, Le Dily S, Vavasseur F, Pavageau A, St Louis EK, Pereon Y, Neunlist M, Derkinderen P, Leclair-Visonneau L. Wake and non-rapid eye movement sleep dysfunction is associated with colonic neuropathology in Parkinson's disease. Sleep. 2024 Mar 11;47(3):zsad310. doi: 10.1093/sleep/zsad310. PMID 38156524